CLINICAL TRIAL: NCT06929468
Title: Cisplatin-induced Cochlear and Vestibular Damage in Head and Neck Squamous Cell Carcinoma: A Cohort Study
Brief Title: Cisplatin-induced Cochlear and Vestibular Damage in Head and Neck Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Simon Jäger (Other)
Collaborators: Klinikum Nürnberg (Other)
Responsible Party: Sponsor-Investigator, Simon Jäger, Head: Institute of Clinical Pharmacology, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Other Study IDs: CPN_PMU002
Record Dates: First submitted 2025-04-07; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Ototoxic Hearing Loss; Ototoxicity, Drug-Induced; Cisplatin-induced Hearing Loss; Cisplatin Ototoxicity; Head and Neck Cancer; Dizzyness; Inner Ear Hearing Loss; Vestibular Disease; Squamous Cell Carcinoma of the Head and Neck; Deafness; Hearing Loss
MeSH Terms: conditions — Ototoxicity; Head and Neck Neoplasms; Dizziness; Hearing Loss, Sensorineural; Vestibular Diseases; Squamous Cell Carcinoma of Head and Neck; Deafness; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Patients can take part in an optional genetic analysis where blood samples will be taken to assess for genes that predispose to developing inner ear damage during chemotherapy with cisplatin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cisplatin chemoradiotherapy: Adult patients with head and neck squamous cell carcinoma receiving cisplatin chemotherapy and radiotherapy.
- Only radiotherapy: Adult patients with head and neck squamous cell carcinoma receiving only radiotherapy.

SUMMARY:
The goal of this observational study is to learn about the occurrence of and to identify suitable strategies for screening and monitoring of inner ear damage in patients receiving cisplatin chemoradiotherapy for head and neck cancer. Researchers will compare patients who are receiving cisplatin chemoradiotherapy to patients who are only receiving radiotherapy. Patients will undergo standardized testing for hearing loss, tinnitus and vestibular dysfunction at baseline, during and after treatment. Optional genetic analyses will aim to identify genes known to predispose to cisplatin-induced ototoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head and neck squamous cell carcinoma
* Cisplatin-based chemoradiotherapy (monotherapy or combination-therapy, adjuvant or neo-adjuvant) or only radiotherapy (control group)
* Age 18 to 85 years
* Signed agreement and willingness to participate in the study and adhere to the study protocol

Exclusion Criteria:

* Severe hearing impairment (WHO grade 3 or 4, corresponding to an audiometric ISO value of ≥61 dB in the better ear at frequencies of 500, 1000, 2000 and 4000 Hz)
* Self-reported tinnitus or vestibular dysfunction in the last 3 months (only lead to exclusion of the corresponding secondary objectives, not to complete exclusion from the study)
* Current cochlear implant
* Concurrent treatment with loop diuretics (e.g. furosemide), aminoglycoside antibiotics or other known ototoxic substances in the last three months
* Acute psychosis or serious psychiatric illness
* Addiction disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck squamous cell carcinoma receiving treatment with cisplatin chemoradiotherapy or only radiotherapy at Klinikum Nuremberg in Nuremberg, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Tinnitus | From enrollment prior to treatment initiation to the last follow-up circa 3 months after completion of treatment.
  Incidence and severity of new or exacerbated tinnitus during treatment with cisplatin chemotherapy measured as impairment according to the Tinnitus Handicap Inventory (THI) score:
  0-16 = no impairment. 18-36 = mild impairment. 38-56 = moderate impairment. 58-76 = severe impairment. 78-100 = catastrophic impairment.
Hearing loss | From enrollment prior to treatment initiation to the last follow-up circa 3 months after treatment completion.
  Incidence of significant hearing loss during treatment with cisplatin chemotherapy described according to CTCAE (Common Terminology Criteria for Adverse Events) in 1-8 kHz audiogram:
  Grade 1 = threshold shift 15-25 dB in 2 contiguous test frequencies in at least one ear.
  Grade 2 = threshold shift >25 dB in 2 contiguous test frequencies in at least one ear.
  Grade 3 = threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear.
  Grade 4 = decrease in hearing to profound bilateral loss, absolute threshold >80 dB at 2 kHz and above.
Vestibular dysfunction | From enrollment prior to treatment initiation to the last follow-up circa 3 months after treatment completion.
  Incidence of dizziness or balance disturbances during treatment with cisplatin chemotherapy as determined through the Dizziness Handicap Inventory (DHI); changes of >18 indicates a clinical relevant worsening in condition:
  0-29 = no to mild impairment. 30-60 = moderate impairment. >60 = severe impairment.

SECONDARY OUTCOMES:
Description of hearing loss through further testing | From enrollment prior to treatment initiation to the last follow-up circa 3 months after treatment completion.
  Description of hearing loss requiring treatment according to the Freiburger Einsilber hearing test (≤80% of speech recognition is an indication for hearing aid): proportion of patients with loss of distortion product otoacoustic emissions (DPOAEs) and new hearing loss in high frequency audiometry at 8 - 16 kHz.
  Investigating the usefulness of high frequency audiometry when compared to DPOAEs for early recognition of ototoxicity.
Description of vestibular damage manifesting as worsening dizzyness or imbalance during treatment with cisplatin | From enrollment prior to treatment initiation to the last follow-up circa 3 months after treatment completion.
  Clinically relevant vestibulopathy: Increase in dizzyness symptoms >18 points on the Dizziness Handicap Inventory (DHI) together with instrumentally measurable pathological changes in vestibular function:
  1. Decrease in VOR-Gain in the video head impulse test (vHIT) (from ca. 1 by 0,2 to 0,8) or new overt or covert saccades.
  2. Decrease in caloric excitability by more than 20%.
  3. Increase in non-elicitable vestibular evoked myogenic potentials (VEMPs) during therapy or a new amplitude asymmetry of more than 50%; prolongation of VEMP latency by more than 0.2 ms.
Description of the incidence and type of cisplatin dose-limiting toxicities | From enrollment prior to treatment initiation to the last follow-up circa 3 months after treatment completion.
  1. Dose-limiting nephrotoxicity, myelosuppression, gastrointestinal side effects (gingival deposits, stomatitis, diarrhoea, severe vomiting), fever, cisplatin-induced polyneuropathy [documented as AESI].
  2. Correlation between median cumulative cisplatin dose and adverse effects.
Assessment of tumour-related quality of life | From enrollment prior to treatment initiation to the last follow-up circa 3 months after treatment completion.
  Completion of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30 + HN43).

OTHER OUTCOMES:
Genetic variants related to cisplatin-induced ototoxicity | Once-off blood sample taken simultaneously with any of the routine blood samples during treatment, can be at any point from study enrollment to the last follow-up visit circa 3 months after treatment completion.
  Prevalence of genetic variants that are predicitve and/or protective of inner ear damage during treatment with cisplatin chemotherapy (optional - patients can choose to only take part in the main study and not in the genetic analysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Nuremberg, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No